CLINICAL TRIAL: NCT04333446
Title: Independent Relationship Between Prealbumin and Circulating Levels of Parathormone Triglycerides and FT3 in Subjects With Overweight or Obesity
Brief Title: Circulating Levels of Pealbumin in Relation to Overweight or Obesity
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Gianluigi Giannelli, Clinical Professor, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: 4/2020
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study was aimed to investigating the relationship between circulating level of prealbumin and parathormone (PTH), triglycerides and triiodothyronine (FT3) in overweight and obese subjects (BMI≥25 Kg/m2)

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI> 25 Kg/m2)

Exclusion Criteria:

* Any kind of drug Hypertension Endocrine diseases (diabetes mellitus, hypo or hyperthyroidism, hypopituitarism, etc.), Chronic inflammatory diseases Renal failure Liver failure Angina pectoris Myocardial infarction and heart failure Genetic heart diseases Thrombocytopenias

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who came to the Outpatient Clinic of Nutrition at the National Institute of Gastroenterology "S. de Bellis," Research Hospital, Castellana Grotte, Italy.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prealbumin | baseline
  Prealbumin (g/L) concentration in serum
Free Triiodothyronine (FT3) | baseline
  FT3 (pg/mL) concentration in serum
Parathormone (PTH) | baseline
  PTH (pg/mL) concentration in serum
Triglycerides | baseline
  Triglycerides (mg/dl) concentration in serum

SECONDARY OUTCOMES:
Height | baseline
  Height in meters
Weight | baseline
  Weight in kilograms
Body mass Index (BMI) | baseline
  BMI (kg/m^2)

CONTACTS AND LOCATIONS:
Locations (1):
- Luisa Lampignano, Castellana Grotte, Italy

IPD SHARING:
Plan to Share IPD: No